CLINICAL TRIAL: NCT05323162
Title: Encapsulated Faecal Microbiota Transplantation to Preserve Residual Beta Cell Function in Patients With Recently-Diagnosed Type 1 Diabetes Mellitus
Brief Title: Encapsulated Faecal Microbiota Transplantation to Preserve Residual Beta Cell Function in Type 1 Diabetes Mellitus
Acronym: ENCAPSULATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nordin Hanssen (Other)
Responsible Party: Sponsor-Investigator, Nordin Hanssen, Internist-endocrinologist, Principial investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL79666.018.21
Record Dates: First submitted 2022-03-17; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Encapsulated autologous fecal microbiota transplantation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Encapsulated autologous fecal microbiota transplantation (Experimental): Encapsulated own microbiota to be transplanted from large- to small intestine by oral ingestion
  Interventions: Other: encapsulated autologous fecal microbiota transplantation

INTERVENTIONS:
Other: encapsulated autologous fecal microbiota transplantation — Individuals will recieve encapsulated freezedried own fecal microbiota to potentially extingish auto-immunity directed against the residual beta cell fraction

SUMMARY:
In this single arm pilot study it will be investigated whether encapsulated autologous fecal microbiota transplantation may be used to halt the decline in residual beta cell function in individuals with recent onset Type 1 diabetes mellitus.

DETAILED DESCRIPTION:
Rationale: The (small) intestinal microbiota composition has been implicated to play an important role in (human) metabolism, as well as autoimmune diseases such as type 1 diabetes mellitus. Faecal microbiota transplantation (FMT) has been shown to significantly alter the microbiota composition, without any serious side effects. It was recently demonstrated that multiple infusions of own faeces (autologous) preserved residual beta cell function up to one year after start of the FMT. Encapsulated autologous FMT provides a safe and feasible option for prolonged treatment on a daily basis, which might stabilize the beta-cell destruction and extend or even bring back the honeymoon period (wherein individuals with recently diagnosed T1D remain wellregulated with minimal doses of insulin).

Objective: confirm the efficacy and feasibility of daily ingested encapsulated freeze-dried autologous (own) faecal matter on the preservation of residual beta cell function as assessed by C-peptide release upon a mixed meal test (MMT) in recently diagnosed type 1 diabetes mellitus (T1D).

Study design: Open label study Study population: Recently diagnosed (0.5-3.5 years of diagnosis) patients with T1D (n=10, aged 18-65 years, BMI 18-30 kg/m2, male/female).

Intervention: After inclusion in the study and a run-in period of 3 months, stools of the participants will be collected and processed into freeze-dried faecal microbiota capsules, which will be ingested daily for 3 months. Participants will be followed for 9 months after inclusion.

Main study parameters/endpoints: The primary endpoint is long-term preservation of beta cell insulin secretion capacity as assessed by stimulated C-peptide AUC0-120min response upon MMT (at -3, 0, 3 and 6 months). The secondary endpoint pertains to changes in plasma biochemistry (HbA1c levels), glucose time-in-range (Freestyle Libre) and subsequent exogenous insulin dose use at -3, 0, 3 and 6 months. The tertiary endpoint is changes in faecal gut microbiota composition at -3, 0, 3 and 6 months, as well as small intestinal microbiota (duodenal biopsy via gastroscopy at 0 and 3 months).

The fourth endpoint is dietary intake and urinary and plasma metabolites at -3, 0, 3 and 6 months.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: This study is considered an intermediate risk study, mainly due to the duodenal biopsies via gastroscopy at 0 and 3 months. 4 MMTs will be performed, for which 70 ml of blood samples will be drawn each visit. The patient will complete several questionnaires, keep track of a food diary and collect urine and faeces prior to study visits. At the study visits BMI and blood pressure will be measured. As of today no adverse events as result of FMT have been reported in this centre. In addition, the use of autologous faeces comes with a lower risk for transmitting any unknown pathogens compared to an allogenic FMT from a lean healthy donor. Moreover, the encapsulated FMT provides an less invasive, well tolerated alternative to the traditional fresh FMT via nasoduodenal tube. As there currently is no therapy to preserve beta cell function in type 1 diabetes, encapsulated autologous FMT can have a potential benefit for the participants

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. Male or female recently diagnosed (0.5-3.5 years) with type 1 diabetes mellitus.
2. Age: 18-65 years
3. BMI: 18-30 kg/m2
4. Remaining residual beta cell function: detectable plasma C-peptide or urinary Cpeptide at inclusion of the study

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. History or symptoms of other autoimmune disease (e.g. hypo- or hyperthyroidism, rheumatoid arthritis).
2. (Expected) prolonged comprised immunity (e.g. due to recent cytotoxic chemotherapy or human immunodeficiency virus (HIV) infection with a CD4 count < 240/mm3).
3. History of a severe disease of the digestive tract, such as celiac disease, chronic diarrhoea (≥3 stools/day for >4 weeks), chronic obstipation (<2 defecations/week for >3 months), Irritable Bowel Syndrome (IBS) (according to Rome IV criteria) or Inflammatory Bowel Disease (IBD).
4. Use of antibiotics, antacid drugs or proton pump inhibitors in the past 3 months or during the study period.
5. Use of pro-/prebiotics in the past three months or during the study period.
6. Smoking or illicit drug use (e.g. MDMA/amphetamine/cocaine/heroin/GHB) in the past three months or use during the study period.
7. Use of >21 units of alcohol per week on average in the past three months.
8. Pregnancy or breast feeding.
9. Inability to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Preservation of residual beta cell insulin secretion capacity | at -3, 0, 3 and 6 months.
  assessed by maximal C-peptide release (residual beta cell function) upon an MMT, AUC0-120 (mmol/ll x min) will be calculated.

SECONDARY OUTCOMES:
HbA1c | At -3, 0, 3 and 6 months.
  Changes in plasma biochemistry HbA1c (mmol/mol)
Glycaemic control | At -3, 0, 3 and 6 months.
  Changes in glucose time in range (% of time during last 14 days) as measured with continuous glucose monitoring device.
Fecal microbiota composition | At -3, 0, 3 and 6 months.
  changes in faecal gut microbiota measured with s16 rRNA sequencing to measure the relative abundance of bacterial microbiota (expressed as relative abundance)
Small intestinal microbiota composition | Fecal: At -3, 0, 3 and 6 months. Duodenal biopsy: 0 and 3 months
  small intestinal microbiota composition measured with s16 rRNA sequencing to measure the relative abundance of bacterial microbiota (in duodenal biopsy), expressed as relative abundance
Questionnaire | At -3, 0, 3 and 6 months.
  validated questionnaires for abdominal complaints (on a 0-5 scale)
Dietary intake | At -3, 0, 3 and 6 months.
  to calculate fiber intake (g/day)

CONTACTS AND LOCATIONS:
Locations (1):
- Academisch Medisch Centrum, Amsterdam, Please Select, Netherlands

IPD SHARING:
Plan to Share IPD: No